CLINICAL TRIAL: NCT02542462
Title: Potential Mechanisms for Intussusception After Rotavirus Vaccine-Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2015-2754
Record Dates: First submitted 2015-06-24; First posted 2015-09-07 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Intussusception; Rotavirus Infections
Keywords: mechanisms for intussusception; rotavirus vaccine
MeSH Terms: conditions — Intussusception; Rotavirus Infections | interventions — RIX4414 vaccine; Rotavirus Vaccines; RotaTeq

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rotarix® alone (Active Comparator): monovalent rotavirus vaccine (Rotarix®, RV1)
  Interventions: Drug: Rotarix®,
- Rotarix®,with other routine vaccines (Active Comparator): monovalent rotavirus vaccine (Rotarix®, RV1), plus additional immunizations
  Interventions: Drug: Rotarix®, with other routine vaccines
- RotaTeq®, alone (Active Comparator): pentavalent rotavirus vaccine (RotaTeq®, RV5)
  Interventions: Drug: RotaTeq®,
- RotaTeq®,with other routine vaccines (Active Comparator): pentavalent rotavirus vaccine (RotaTeq®,RV5) plus additional immunizations
  Interventions: Drug: RotaTeq®, with other routine vaccines

INTERVENTIONS:
Drug: Rotarix®, — Single oral dose of licensed rotavirus vaccine given alone
  Other Names: Rotavirus vaccine
  Arms: Rotarix® alone
Drug: Rotarix®, with other routine vaccines — Single oral dose of licensed rotavirus vaccine given with other routine vaccines
  Other Names: Rotavirus vaccine
  Arms: Rotarix®,with other routine vaccines
Drug: RotaTeq®, — Single oral dose of licensed rotavirus vaccine given alone
  Other Names: Rotavirus vaccine
  Arms: RotaTeq®, alone
Drug: RotaTeq®, with other routine vaccines — Single oral dose of licensed rotavirus vaccine given with other routine vaccines
  Other Names: Rotavirus vaccine
  Arms: RotaTeq®,with other routine vaccines

SUMMARY:
This is a prospective randomized clinical trial that aims to evaluate the potential effects of the first dose of rotavirus vaccines on gastrointestinal motility and anatomy and blood and stool cytokine responses. It will also assess the association between these outcomes and the pattern of the shedding of vaccine strain rotavirus in the stool. Infants will be randomized to one of four arms: monovalent rotavirus vaccine (Rotarix®, RV1) alone, RV1 with other recommended vaccines, pentavalent rotavirus vaccine (RotaTeq®, RV5) alone, or RV5 with other recommended vaccines. Data derived from the pilot study will be used to assess the feasibility of conducting a larger scale study.

DETAILED DESCRIPTION:
Healthy infants 6-13 weeks of age will be randomized (1:1:1:1) to receive either, RV1 alone, RV1 with Advisory Committee on Immunization Practices (ACIP) routinely recommended immunizations (Diphtheria, Tetanus and Pertussis (DTaP), Haemophilus influenza type b (Hib), pneumococcal conjugate (PCV13), Hepatitis B (HBV) and inactivated polio (IPV)), RV5 alone or RV5 with ACIP routinely recommended immunizations. Imaging study personnel and parents will be blinded to the rotavirus vaccine type; parents will be informed about the rotavirus vaccine type at the completion of the study. Up to 100 infants will be enrolled.

Recruitment and enrollment will occur prior to the first clinic visit. There will be four study visits including the recruitment/enrollment visit and three clinic visits. Infants will be randomized to either RV1, RV1 plus other immunizations, RV5 alone, or RV5 plus other immunizations. Clinic Visit 1 (day 0) will include blood, saliva, stool and breast milk collection . The MRI and ultrasound will be performed prior to vaccination. Children will receive the immunizations to which they are randomized. Imaging personnel and parents will be blinded to rotavirus vaccine type; they will be informed about other vaccines administered. A second MRI and ultrasound will be performed at Clinic Visit 2 (day 5) and blood and stool samples collected. Parents will be unblinded at the completion of Clinic Visit 3 (day 14). Arrangements will be made to get remaining doses of same rotavirus vaccine. Daily stool samples will be collected at home during the 15 day study period (on vaccination day 0 and for next 14 days). A memory aid will be completed to collect reactogenicity data on days 0 and for the next 14 days. Remaining stools and reactogenicity data from parents will be collected at Visit 3.

The investigators will assess blood and stool cytokine responses and intestinal anatomy and motility after rotavirus vaccination by comparing pre-vaccination with post-vaccination responses in the study infants. Cytokines and intestinal anatomy and motility will be assessed at baseline (Visit 1, the day of vaccine receipt) and 5 days after vaccination (Visit 2). For both blood and stool, the following cytokines will be tested: IL-2, IL-6, IL-7, IL-8, IL-15, INF-γ and TNF-α. Additional biomarkers may be studied.

ELIGIBILITY:
Inclusion Criteria:

1. healthy infant 6 to 13 weeks (12 weeks and 6 days) of age at day of rotavirus vaccine administration
2. free of obvious health problems as established by medical history and confirmed with infant's primary physician prior to Visit 1
3. parent/legal guardian willing to have infant feed from a bottle for contrast
4. parent/legal guardian willing and capable of signing informed consent
5. parent/legal guardian and infant expected to be available for entire study
6. parent/legal guardian can be reached by telephone
7. parent/legal guardian expresses willingness to complete study procedures and receive 2 month immunizations, according to recommended schedule

Exclusion Criteria:

1. gestational age of <37 weeks
2. infant unable to fast for 4 hours prior to MRI procedure
3. receipt of any vaccine except initial HBV (must have at least 28 days between HBV and Visit 1 to be included)
4. history of severe allergic reaction to HBV vaccine
5. contraindications for any of the routine vaccines

   1. Severe Combined Immune Deficiency
   2. history of intussusception
6. precautions for either RV1 or RV5 (may interfere with study outcomes)

   a. altered immunocompetence i. infants with primary and acquired immunodeficiency states, cellular immunodeficiency, hypogammaglobulinemic and dysgammaglobulinemic states ii. infants with blood dyscrasias, leukemia, lymphomas, or other malignant neoplasms affecting the bone marrow or lymphatic system iii. infants on immunosuppressive therapy (including high-dose systemic corticosteroids) iv. infants who are HIV-exposed or infected b. acute gastroenteritis c. moderate or severe acute illness with or without fever d. pre-existing chronic gastrointestinal diseases (e.g., congenital malabsorption syndromes, Hirschsprung's disease, or short-gut syndrome) e. infants with spina bifida or bladder exstrophy (latex rubber is contained in the RV1 oral applicator)
7. sensitivity to latex (latex rubber is contained in the RV1 oral applicator)
8. febrile illness within previous 14 days (axillary temperature of 100.4◦ F or higher)
9. history of vomiting (forceful expulsion of partially digested milk/food) and/or diarrhea (3 watery stools) within 14 days of Visit 1
10. receipt of any steroids, immunoglobulins, other blood products/transfusion
11. receipt of non-steroidal anti-inflammatory drugs in previous 72 hours (may affect cytokine response)
12. receipt of an antipyretic medication (acetaminophen or ibuprofen) within 72 hours prior to the first dose of rotavirus vaccine or is already planning to administer a prophylactic antipyretic medication on the day of and the day following vaccination (this exclusion does not apply if the caretaker indicates he/she might administer antipyretics after vaccination to reduce a fever)
13. is enrolled or plans to enroll in another clinical trial with an investigational product while participating in this study (observational studies are allowed)
14. any condition which, in the opinion of the investigators, may post a health risk to the subject or interfere with the MRI or vaccine evaluation
15. currently receiving medication for gastroesophageal reflux (GERD) or any other gastrointestinal condition including colic
16. infant who is a relative of any research study personnel
17. allergy to barium
18. failed newborn hearing screening

    -

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A. Staat, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Karen Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Cincinnati Children's Hosptital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period, there were 252 children screened and of these, 238 were eligible for enrollment. These subjects were identified through screening at a primary care clinic and through advertisement
Pre-assignment Details: 43 of 144 enrolled participants withdrew prior to randomization
Period: Overall Study
Arm/Group | Rotarix® Alone | Rotarix®,With Other Routine Vaccines | RotaTeq®, Alone | RotaTeq®,With Other Routine Vaccines
Started | 25 | 25 | 25 | 26
Completed | 25 | 25 | 25 | 25
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix® Alone | Rotarix®,With Other Routine Vaccines | RotaTeq®, Alone | RotaTeq®,With Other Routine Vaccines | Total
Number analyzed (Participants) | 25 | 25 | 25 | 26 | 101
Age, Continuous [Mean (Full Range); unit: weeks] | 8.5 [6 to 10.6] | 8 [6 to 10.7] | 8.2 [6.1 to 10.1] | 8.4 [6.1 to 10.4] | 8.2 [6 to 10.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 13 | 12 | 45
  Male | 13 | 17 | 12 | 14 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 23 | 25 | 24 | 26 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 21 | 23 | 21 | 23 | 88
  White | 1 | 0 | 3 | 3 | 7
  More than one race | 3 | 2 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 25 | 26 | 101
Gestational age at birth (weeks) [Mean (Full Range); unit: weeks] | 38.6 [37 to 41] | 38.8 [37 to 41] | 38.9 [37 to 42] | 38.8 [37 to 41] | 38.8 [37 to 42]
Birthweight [Mean (Full Range); unit: kilograms] | 3 [1.8 to 3.7] | 3 [1.9 to 3.7] | 3 [1.8 to 4.1] | 3 [2.3 to 3.7] | 3 [1.8 to 4.1]

OUTCOME MEASURES:

1. Primary Outcome: The Effects of RV1 and RV5 With or Without Other Routine Immunizations on Gastrointestinal Anatomy
Description: Number of subjects with an increase in the number of abdominal lymph nodes, as measured by abdominal ultrasound, or an increase of 1 mm or more of terminal ileum wall thickness, as measured by abdominal MRI, from Day 0 (Visit 1) to Day 4-6 (Visit 2)
Time Frame: 4- 6 days
Population: Subjects had an abdominal MRI followed by an abdominal ultrasound prior to receiving vaccines at Day 0 (Visit 1). They returned 4-6 days later for follow up MRI and Ultrasound post vaccination (Visit 2) Terminal ileum thickness was measured and compared pre-post. Abdominal lymph nodes seen on ultrasound were compared pre-post
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix® Alone | Rotarix®,With Other Routine Vaccines | RotaTeq®, Alone | RotaTeq®,With Other Routine Vaccines
Number analyzed (Participants) | 25 | 25 | 25 | 25
Participants
  Terminal Ileum increase | 2 | 1 | 0 | 1
  Lymph node increase | 11 | 9 | 5 | 10
Statistical Analysis 1: Comparison: Rotarix® Alone vs Rotarix®,With Other Routine Vaccines vs RotaTeq®, Alone vs RotaTeq®,With Other Routine Vaccines; The test is to see a difference among the four groups and the pre to post change of the primary outcomes; Test type: Superiority; p = 0.2, Fisher Exact — P value for the number of subjects with an increase of 1 mm or more of terminal ileum from pre to post was 0.2
Statistical Analysis 2: Comparison: Rotarix® Alone vs Rotarix®,With Other Routine Vaccines vs RotaTeq®, Alone vs RotaTeq®,With Other Routine Vaccines; The test is to see a difference among the four groups and the pre to post change of the primary outcomes; Test type: Superiority; p = 0.3, Fisher Exact — P value for change in the number of subjects with an increase in number of lymph nodes from pre to post was 0.3

2. Primary Outcome: The Feasibility of Conducting a Larger Scale Study as Determined by Study Recruitment Rates (Number of Participants Eligible/Participants Who Enrolled)
Description: Study will be determined to be feasible on a larger scale if 10% or more of eligible subjects enroll in the study
Time Frame: 15 months
Population: During the study period, there were 252 children screened and of these, 238 were eligible for enrollment. These subjects were identified through screening at a primary care clinic and through advertisement.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Infants were randomized to one of four arms: monovalent rotavirus vaccine (Rotarix(r) RV1) alone, RV1 with other recommended vaccines, pentavalent rotavirus vaccine (RotaTeq(r) RV5) alone, or RV5 with other recommended vaccines
Arm/Group | All Study Participants
Number analyzed (Participants) | 238
Participants | 144

3. Primary Outcome: The Feasibility of Conducting a Larger Scale Study as Determined by the Percentage of Participants Who Completed All Study Visits
Description: Study will be determined to be feasible on a larger scale if 70% or more of randomized subjects complete all study visits and remain in the study until completion
Time Frame: 15 months
Population: All randomized subjects, irrespective of arm assignment
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 101
Participants | 100

ADVERSE EVENTS:
Time Frame: 15 days
Description: solicited adverse events included fever, diarrhea, vomiting, irritability and hematochezia. Parents of infants filled out a memory aid for 15 days recording any of these events.
Arm/Group | Rotarix® Alone | Rotarix®,With Other Routine Vaccines | RotaTeq®, Alone | RotaTeq®,With Other Routine Vaccines
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25 | 25/25 | 25/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotarix® Alone (N=25) | Rotarix®,With Other Routine Vaccines (N=25) | RotaTeq®, Alone (N=25) | RotaTeq®,With Other Routine Vaccines (N=26)
Fever (Infections and infestations) | 4 (4) | 1 (1) | 6 (6) | 1 (1) — Axillary temperature equal or greater to 99.5 Fahrenheit
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2) — Three looser than normal stools a day
Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (7) | 5 (5) | 8 (8) — One episode of vomiting
Irritability (Nervous system disorders) | 17 (17) | 15 (15) | 13 (13) | 16 (16) — Crying more than usual

LIMITATIONS AND CAVEATS:
This was a pilot study to assess the feasibility of conducting the outlined study and was not powered to detect differences in the anatomy pre-versus post immunization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT02542462/Prot_SAP_000.pdf